CLINICAL TRIAL: NCT04429438
Title: Primary, Booster and Consolidation Multi-CAR-T Cell Therapy for the Treatment of Refractory B Cell Lymphomas
Brief Title: Multi-CAR-T Cells Targeting B Cell Lymphomas
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: The Seventh Affiliated Hospital of Sun Yat-sen University (Other); Shenzhen Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-20006
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: B Cell Lymphoma (BCL)
Keywords: CAR-T; CD19; CD20; CD22; CD70; PSMA; CD13; CD79b; GD2; PMBCL; CNS-BCL
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4SCAR19 and 4SCAR20/22/70/PSMA/13/79b/GD2 (Experimental): Patients who have relapsed and refractory B cell lymphoma (BCL) after chemotherapy will be treated with a combination of 4SCAR gene-engineered T cells.
  Interventions: Biological: 4SCAR19 and 4SCAR20/22/70/PSMA/13/79b/GD2

INTERVENTIONS:
Biological: 4SCAR19 and 4SCAR20/22/70/PSMA/13/79b/GD2 — Patients who have relapsed and refractory B cell lymphoma (BCL) after conventional chemotherapy will be treated with multiple 4SCAR gene-engineered T cells

SUMMARY:
This study aims to evaluate safety and efficacy of a combination of 4th generation chimeric antigen receptor gene-modified T cells targeting B cell surface molecules including CD19 and alternative CARTs as booster and consolidation treatment for patients with highly resistant B cell lymphomas, including primary mediastinal B cell lymphoma (PMBCL) and BCL involving central nervous system (CNS-BCL). Clinical response and development of a simplified and standardized lentiviral vector and cell production protocol will be investigated. This is a phase I/II trial enrolling patients from multiple clinical centers.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR) T cell therapy has proven effective in treating B cell malignancies. However, post CD19-CART relapses occur at high rate due to the CD19 antigen loss or the exhaustion of CART cells. Furthermore, the success of treating relapsed/refractory B cell lymphoma (BCL) such as primary mediastinal B-cell lymphoma (PMBCL) and CNS-involved BCL has been limited. To overcome tumor escape and prolong in vivo CART efficacy, we have developed a novel multiple CAR-T therapy regimen including booster and consolidation CART applications to to target highly-refractory cancer. Selected patients will be enrolled after target antigen confirmation including CD19, CD20, CD22, CD70, CD13, CD79b, GD2 and PSMA through immunostaining of their tumor specimens. The aim is to evaluate safety and long term efficacy of the multiple CART therapy strategy in the BCL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 6 months.
2. Primary B cell lymphoma surface expression of CD19 and/or CD22/CD70/PSMA/ CD13/CD79b/GD2 molecules.
3. The KPS score over 80 points, and survival time is more than 1 month.
4. Greater than Hgb 80 g/L.
5. No contraindications to blood cell collection.

Exclusion Criteria:

1. Accompanied with other active diseases, and difficult to assess response after treatment.
2. Bacterial, fungal, or viral infection, unable to control.
3. Living with HIV.
4. Active HBV and HCV infection.
5. Pregnant and nursing mothers.6. under systemic steroid treatment within a week of the treatment.

7. Prior failed CAR-T treatment.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of fourth generation anti-CD19 and anti-CD20/CD22/CD70/PSMA/CD13/CD79b/GD2 CAR-T cells infusion | 24 weeks
  Safety of fourth generation anti-CD19 and anti-CD20/CD22/CD70/PSMA/CD13/CD79b/GD2 CAR-T cells in patients with relapsed B cell lymphoma (BCL) using CTCAE 4 standard to evaluate the level of adverse events

SECONDARY OUTCOMES:
Anti tumor activity of fourth generation anti-CD19 and anti-CD20/CD22/CD70/PSMA/CD13/CD79b/GD2 CAR-T cells infusion | 1 year
  Objective responses (complete response (CR) + partial response (PR)) are assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Shenzhen Geno-Immune Medical Institute, Shenzhen, Guangdong
  - The Seventh Affilliated Hospital, Sun Yat-Sen University, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No